CLINICAL TRIAL: NCT00668382
Title: Phase I Study To Evaluate The Toxicity And Feasibility Of Intra-Tumoral Injection Of Alpha-Gal Glycosphingolipids In Patients With Advanced Or Refractory Solid Tumors
Brief Title: Evaluate The Toxicity And Feasibility Of Intra-Tumoral Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Giles Whalen, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UM200702
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Neoplasm Metastases
Keywords: Cancerous solid tumors; Alpha-Gal Glycosphingolipids
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alpha-Gal Glycosphingolipid injection (Experimental): Intervention: Intratumoral injection of a single dose of Alpha-Gal Glycosphingolipid (0.1 mg,1mg, 10mg)
  Interventions: Biological: Alpha-Gal Glycosphingolipid

INTERVENTIONS:
Biological: Alpha-Gal Glycosphingolipid — Intra-tumoral injection of Alpha-Gal Glycosphingolipid to evaluate toxicity

SUMMARY:
This is a Phase I pilot study to evaluate the toxicity and feasibility of intratumoral injection (Glycosphingolipids) GSL alpha-GAL (beta-galactosidase) in patients with advanced, refractory solid tumors who have failed standard therapies or are not eligible for standard treatment.

DETAILED DESCRIPTION:
Intratumoral injection of alpha gal glycolipid in experimental knockout mouse model systems incorporates into tumor cell membranes and presents these xeno-transplantation epitopes to antigen presenting cells with that particular tumor's tumor associated antigens (TAA). Thus this maneuver converts any individual tumor into an in situ tumor vaccine without the need to isolate, purify or supply TAA exogenously. The effects in these model systems demonstrate both the upregulation of cytotoxic T cells which react against the particular tumor's TAA, as well as resolution of injected primary tumor and eradication and prevention of metastatic disease at distant sites. This current study was undertaken to investigate the safety and feasibility of such an approach in humans. The major toxicity concerns are acute allergic or complement activation reactions or development of autoimmunity. The primary treatment is a single intratumoral injection of alpha gal glycolipid. The study design is a standard dose escalation design and the primary endpoint is Dose limiting toxicity at one month after injection (grade 3 or 4. Subjects are followed until death utilizing standard clinical imaging and evaluation to judge overall tumor response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with solid tumors who have failed standard therapies, or are not candidates for standard therapies.
2. Patients must have at least one measurable lesion that is accessible and suitable for injection of the GSL alpha-GAL.
3. Patients should not be undergoing any active treatment with chemotherapy, radiotherapy, or steroids (either because the patient or the treating physician have decided not to employ these therapies at this time, or because they had already been tried and failed). If they have been treated with these modalities, the treatments should have been completed at least two weeks prior to date of injection of GSL alpha-GAL.
4. Patients should be judged by the investigator to be able to undergo safely the procedure needed to inject the tumor with GSL alpha-GAL.
5. Age equal or over 18 years old.
6. ECOG (Eastern Cooperative Oncology Group ) performance of less than 2. (International Normalized Ratio) INR less than 1.5 and a (Partial Thromboplastin Time) PTT no greater than normal limits within 1 week prior to intra-tumoral injection (For patients who requires invasive procedure for intra-tumoral injection).
7. Laboratory Criteria (completed equal or less 2 weeks before enrollment) Hematologic: (White Blood Cell Count) WBC equal or above 3500/millimeter-cubed or (Absolute Neutrophil Count) ANC equal or above 1500/millimeter-cubed and platelet count equal or above 100,000/ millimeter-cubed.

   Hepatic: Total bilirubin equal or less 4.0 milligrams/deciliter. Renal: Creatinine equal or less 2.2 milligrams/deciliter.
8. Patients must be negative for HIV (circulating antibody), Hepatitis B (circulating antigen), and Hepatitis C (circulating antibody).
9. Patients should have an expected survival of more than 6 weeks and should not have other systemic anti-tumor treatments planned during this time frame.

Exclusion Criteria:

1. Patients who are pregnant (as determined by a positive serum HCG (Human Chorionic Gonadotropin) in patients of childbearing potential) or nursing.
2. Patients under the age of 18.
3. Patients with severe infections or septicemia.
4. Patients with a history of autoimmune disease.
5. Patients in, or about to be in, active treatment with chemotherapy or steroids.
6. Patients who refuse HIV/hepatitis testing and patients who do not sign an approved consent form.
7. Patient has received other investigational drugs within 14 days before enrollment or is expected to participate in an experimental drug study during this study treatment.
8. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giles Whalen, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Lugade AA, Moran JP, Gerber SA, Rose RC, Frelinger JG, Lord EM. Local radiation therapy of B16 melanoma tumors increases the generation of tumor antigen-specific effector cells that traffic to the tumor. J Immunol. 2005 Jun 15;174(12):7516-23. doi: 10.4049/jimmunol.174.12.7516. PMID 15944250
- [Result] Malmberg KJ. Effective immunotherapy against cancer: a question of overcoming immune suppression and immune escape? Cancer Immunol Immunother. 2004 Oct;53(10):879-92. doi: 10.1007/s00262-004-0577-x. Epub 2004 Jul 28. PMID 15338206
- [Result] DiGiacomo A, North RJ. T cell suppressors of antitumor immunity. The production of Ly-1-,2+ suppressors of delayed sensitivity precedes the production of suppressors of protective immunity. J Exp Med. 1986 Oct 1;164(4):1179-92. doi: 10.1084/jem.164.4.1179. PMID 2944983
- [Result] Shimizu J, Yamazaki S, Sakaguchi S. Induction of tumor immunity by removing CD25+CD4+ T cells: a common basis between tumor immunity and autoimmunity. J Immunol. 1999 Nov 15;163(10):5211-8. PMID 10553041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from medical and surgical oncology clinics with currently untreatable tumors from march 2007 through June 2011
Pre-assignment Details: No assignment to separate arms, Patients had to be off any active treatment for their advanced tumors for at least 2 weeks before entry onto study and a month after. Two subjects withdrew after screening and consent because of stroke (1) and insurance refusal(1). Two patients dropped out in the first month due to treatment needs.
Period: Overall Study
Arm/Group | Alpha-Gal Glycosphingolipid Injection
Started | 11 (beginning of trial)
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alpha-Gal Glycosphingolipid Injection
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Greater Than Grade 3 or 4 Toxicity
Description: Grade 3/4 Toxicity occurring in a participant within a month of intratumoral injection
Time Frame: 1 month
Population: Dose escalating Phase 1 scheme: three participants for each dose cohort. The second patient in the last (10 mg) dose cohort developed and adverse event (infection at injection site) and so three more participants were entered and analyzed at that dose
Measure: Number; unit: participants
Groups:
- Intratumoral Injection: Single Intratumoral injection of Alpha Gal Glycosphingolipid. Three dose cohorts (0.1mg, 1mg, 10mg)
Arm/Group | Intratumoral Injection
Number analyzed (Participants) | 11
participants | 1

ADVERSE EVENTS:
Time Frame: Over one month
Description: patients followed for as long as they lived per clinical care protocols
Arm/Group | Intratumoral Injection
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intratumoral Injection (N=11)
surgical site infection (Surgical and medical procedures) | 1 (1) — Patient developed an abscess (UGI flora) at an injection site in the pancreatic body one week after injection via an EUS guided approach. This required hospitalization, IV antibiotics and drains placed by interventional radiology. Subject recovered.

LIMITATIONS AND CAVEATS:
No allergic/immune toxicity. The single toxicity/AE was bacterial infection with UGI flora at injection site following EUS (endoscopic ultra-sound) guided injection of pancreatic cancer. Added injections covered with antibiotic prophylaxis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes